CLINICAL TRIAL: NCT00800267
Title: A 6-month, Randomized, Double-masked Comparison of Fixed Combination of Latanoprost and Timolol With the Individual Components, Continuing Into a 6-month Open Label Safety Study of Fixed Combination in Patients With Glaucoma or Ocular Hypertension. A Multicenter Study in the United States
Brief Title: A Study of Glaucoma or Ocular Hypertension in Patients Within the United States
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96TIPG005; A6641006
Record Dates: First submitted 2008-11-03; First posted 2008-12-02 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2009-03

CONDITIONS: Ocular Hypertension; Glaucoma
Keywords: glaucoma; ocular hypertension; Fixed combination latanoprost-timolol; latanoprost; timolol
MeSH Terms: conditions — Ocular Hypertension; Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fixed combination of latanoprost 0.005% and timolol 0.5% (Experimental)
  Interventions: Drug: fixed combination latanoprost-timolol
- latanoprost 0.005% (Active Comparator)
  Interventions: Drug: latanoprost 0.005%
- Timolol - 0.5% (Active Comparator)
  Interventions: Drug: timolol 0.5%

INTERVENTIONS:
Drug: latanoprost 0.005% — placebo in the morning and latanoprost .005% in the evening
  Arms: latanoprost 0.005%
Drug: fixed combination latanoprost-timolol — one drop in the morning and placebo in the evening
  Arms: Fixed combination of latanoprost 0.005% and timolol 0.5%
Drug: timolol 0.5% — one drop in the morning and evening
  Arms: Timolol - 0.5%

SUMMARY:
Safety and efficacy study comparing between fixed combination latanoprost-timolol and its component parts.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral primary open angle glaucoma, capsular glaucoma, pigmentary glaucoma or ocular hypertension.
* Patients currently on IOP reducing therapy: IOP greater than or equal to 25mmHg (Ltwo IOP determinations at pre-study separated by at least one hour) OR Patients without IOP reducing therapy: IOP greater than or equal to 30mmHg (two IOP determinations at pre-study separated by at least one hour).

Exclusion Criteria:

* History of acute angle closure or closed/barely open anterior chamber angle.
* Current use of contact lenses.
* Ocular surgery or argon laser trabeculoplasty (ALT) within three months prior to pre-study visit.
* Ocular inflammation/infection occurring within three months prior to pre-study visit.
* Hypersensitivity to benzalkonium chloride or to any other component of the study drug solutions.
* Other abnormal ocular condition or symptom preventing the patient from entering the study, according to the investigator's judgement.
* Patients with conditions in which treatment with B-blocking agents are contraindicated: cardiac failure, sinus bradycardia, second and third degree atrio-ventricular block.
* Patients with conditions in which treatment with B-blocking agents are contraindicated: bronchial asthma, history of bronchial asthma or chronic obstructive pulmonary disease.
* Inability to adhere to treatment/visit plan.
* Have participated in any other clinical study within one month prior to pre-study visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 1997-07; Primary Completion 1999-06 (Actual); Study Completion 1999-06 (Actual)

PRIMARY OUTCOMES:
The differences from baseline in diurnal IOP reduction after six months of treatment will be tested between the fixed combination and the monotherapy groups. | 6 months
Primary objective: to demonstrate that the fixed combination of latanoprost and timolol has a better IOP-reducing effect than the individual monotherapies. | 6 months

SECONDARY OUTCOMES:
To examine, within treatment groups, the diurnal IOP reducing effect from baseline for all effect from baseline between the monotherapies latanoprost and timolol | 6 months
To compare the diurnal IOP reducing effect from baseline between the monotherapies latanoprost and timolol at Week 26 | 6 months
To compared the number of treatment failures and patients withdrawn due to uncontrolled IOP from baseline to Week 26 between treatment groups | 6 months
To describe the IOP development from baseline to Week 26 for all treatment groups | 6 months
To compared the IOP reducing effect from baseline to Week 26 of the monotherapies with the IOP reducing effect from Week 26 to Week 52 of the fixed combination | 6 months
To examine, within the fixed combination treatment group, the diurnal IOP reducing effect from baseline to Week 26 and Week 52 | 6 months
To follow the safety variables throughout the study periods. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- United States (42):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Largo, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, East Point, Georgia
  - Pfizer Investigational Site, Griffin, Georgia
  - Pfizer Investigational Site, Morrow, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Wheaton, Illinois
  - Pfizer Investigational Site, Elkhart, Indiana
  - Pfizer Investigational Site, Mishawaka, Indiana
  - Pfizer Investigational Site, South Bend, Indiana
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Owings Mills, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Golden Valley, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Warrensburg, Missouri
  - Pfizer Investigational Site, Concord, New Hampshire
  - Pfizer Investigational Site, South Plainfield, New Jersey
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Matthews, North Carolina
  - Pfizer Investigational Site, Monroe, North Carolina
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Wyomissing, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Galveston, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=96TIPG005&StudyName=A%20study%20of%20glaucoma%20or%20ocular%20hypertension%20in%20patients%20within%20the%20United%20States.